CLINICAL TRIAL: NCT04594486
Title: Long Term Results of Medical Treatment for Acute Appendicitis
Brief Title: Medical Treatment for Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Barış Sevinç, Assoc. Prof., Uşak University
Other Study IDs: app001
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Medical treatment of acute appendicitis — All cases will be treated medically and will be followed for recurrences

SUMMARY:
Medical treatment for acute appendicitis

DETAILED DESCRIPTION:
Patients with clinically and radiologically approved acute appendicitis will be treated medically. The main aim of the study is to define the long term results of medical treatment for acute appendicitis. Patients will be followed by clinical visits and recurrences will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* clinically and radiologically approved acute appendicitis
* approved and signed the informed consent form

Exclusion Criteria:

* perforated cases
* cases with peritonitis
* patient wish for surgical treatment
* allergy to drugs used in medical treatment of acute appendicitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute appendicitis
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
recuurence | 5 years
  recuurent acute appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: Barış Sevinç, M.D., Principal Investigator — Uşak University Medical School
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided